CLINICAL TRIAL: NCT05056337
Title: Efficacy and Safety of Toripalimab in Combination With Lenvatinib and TACE for Conversion Therapy in Patients With Potentially Resectable Hepatocellular Carcinoma: a Prospective, Multicenter, Randomized Controlled Study
Brief Title: Toripalimab in Combination With Lenvatinib and TACE for Conversion Therapy in Patients With Potentially Resectable HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-338(2)
Record Dates: First submitted 2021-08-17; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Toripalimab; Lenvatinib; TACE; conversion therapy; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients with potentially resectable HCC who meet the study inclusion criteria will be treated with lenvatinib(8mg/d for BW<60kg and 12mg for BW≥60kg) in combination with toripalimab(240mg iv Q3W) and TACE (on demand). Tumor response will be regularly evaluated, data will be collected, and complete surgical resection will be evaluated by an independent review committee, the conversion resection rate will be calculated, and patient survival will be assessed.
  Interventions: Drug: Lenvatinib 4 MG Oral Capsule [Lenvima]; Drug: Toripalimab; Procedure: TACE
- Control group (Active Comparator): Patients with potentially resectable HCC who meet the study inclusion criteria will be treated with TACE alone. Tumor response will be regularly evaluated, data will be collected, and complete surgical resection will be evaluated by an independent review committee, the translational resection rate will be calculated, and patient survival will be assessed.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib 4 MG Oral Capsule [Lenvima] — patients will be treated with lenvatinib in combination with toripalimab and TACE (on demand)
  Arms: Treatment group
Drug: Toripalimab — patients will be treated with lenvatinib in combination with toripalimab and TACE (on demand)
  Arms: Treatment group
Procedure: TACE — Hepatic arterial chemoembolization

SUMMARY:
Study introduction: this is a multicenter, randomized controlled study of patients with histopathologically confirmed hepatocellular carcinoma (HCC) who have not previously received systematic treatment for HCC, all the patients are Chinese stage IIb/IIIa (BCLC stage B/C), and have not developed extrahepatic metastases. Follow-up, data collection and analysis will be performed for patients who meet the study inclusion criteria and will be treated with lenvatinib plus toripalimab and TACE (on demand) or TACE alone, so as to compare the objective response rate (ORR), overall survival (OS), progression-free survival (PFS), ratio of conversion resection, and safety between the two cohorts.

DETAILED DESCRIPTION:
The study includes two groups:

Treatment group: patients with potentially resectable HCC who meet the study inclusion criteria will be treated with lenvatinib in combination with toripalimab and TACE (on demand). Tumor response will be regularly evaluated, data will be collected, and complete surgical resection will be evaluated by an independent review committee, the conversion resection rate will be calculated, and patient survival will be assessed.

Control group: patients with potentially resectable HCC who meet the study inclusion criteria will be treated with TACE. Tumor response will be regularly evaluated, data will be collected, and complete surgical resection will be evaluated by an independent review committee, the translational resection rate will be calculated, and patient survival will be assessed.

The maximum duration of study treatment for each subject is expected to be 48 weeks, with efficacy evaluation by the MDT after 2 TACE treatments to determine whether subjects meet the surgical criteria.

This study is a multicenter, randomized controlled study. The primary endpoint is the objective response rate (ORR). Historical data showed that the objective response rate of patients in the TACE group was about 40%. The objective response rate of lenvatinib in combination with toripalimab and TACE is expected to reach 60%. Using a two-sided Z test of pooled variance, α is set to 0.05, power is set to 0.8, and patients will be assigned at a 1:1 ratio. The required sample sizes are 98 (treatment group) and 98 (control group), and a total of 220 subjects are planned to be prospectively observed, taking into account a dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of 18-75 years old;
2. Clinical or histopathological diagnosis of hepatocellular carcinoma;
3. ECOG PS score of 0-1, Child-Pugh grade A;
4. Chinese stage IIb/IIIa (equal to BCLC B/C) patients with portal vein tumor thrombus (according to the Japanese PVTT grading criteria Vp3-Vp4) or more than 3 tumor nodules, without extrahepatic metastasis;
5. According to the evaluation by the site multi-disciplinary team (MDT), surgical resection is not the current preferred treatment;
6. No previous systemic treatment for hepatocellular carcinoma; no previous use of PD-1 inhibitor, PD-L1 inhibitor, lenvatinib or sorafenib;
7. Previous TACE treatment for 0-2 times
8. The patients in the treatment group voluntarily and have decided to receive treatment of lenvatinib in combination with toripalimab and TACE, and sign an informed consent form. Additional identification of qualified subjects: subjects who have received at least one combination medication enter the safety evaluation; subjects who have received at least one imaging evaluation after treatment enter the efficacy evaluation. The patients in the control group treated with TACE alone have at least one imaging evaluation.
9. Patients with HBV infection (characterized by hepatitis B surface antigen [HBsAg] positive and/or hepatitis B core antibody [anti-HBcAb], with detectable HBV DNA [>10 IU/mL]) should be treated with antiviral therapy according to clinical routine, so as to ensure adequate viral suppression (HBV DNA≤2000 IU/mL or 104) before enrollment. Patients must maintain antiviral therapy during the study period and within 6 months after the last study drug administration; patients with positive hepatitis B core antibody (HBc) and undetectable HBV DNA (<10 IU/mL) will be not required to receive antiviral therapy before enrollment; these patients will be checked every cycle to monitor HBV DNA levels; if HBV DNA is detected (> 10 IU/mL), antiviral therapy will be initiated; patients with detectable HBV DNA must continue to receive antiviral therapy during the study

Exclusion Criteria:

1. Clinical or pathological diagnosis of mixed liver cancer, fibrolamellar hepatocellular carcinoma or other non-hepatocellular malignant tumor components;
2. Hematological examination: PLT<50×109/L, WBC<3.0×109/L or not meet the requirements of TACE treatment;
3. Coagulation function: international normalized (prothrombin time) ratio (INR) > 1.2;
4. Liver function indicators: serum albumin (ALB) < 2.8 g/dl, serum total bilirubin (TBIL) > 1.5 times the upper limit of normal (excluding those with biliary obstruction), serum transaminase (ALT and AST) > 3 times the upper limit of normal;
5. Renal function indicators: serum creatinine (CR) > 1.5 times the upper limit of normal;
6. Uncontrollable hypertension (defined as diastolic blood pressure > 90 mmHg or systolic blood pressure > 150 mmHg);
7. Patients with bile duct tumor thrombi, superior mesenteric vein tumor thrombi and diffuse portal vein tumor thrombi;
8. Participated in other clinical trials 30 days before screening;
9. Accompanied by hepatic encephalopathy, Gilbert syndrome, sclerosing cholangitis, etc.;
10. Acute gastrointestinal bleeding recorded within the last 3 months;
11. Have a history of allogeneic transplantation (such as liver transplantation);
12. Patients with acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV) DNA > 2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA > 103 copies/ml; those who are positive for both hepatitis B surface antigen (HbsAg) and anti-HCV antibodies.
13. Patients who have autoimmune diseases or a history of autoimmune diseases or syndromes requiring systemic use of steroids / immunosuppressants, including hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism etc.
14. Be suspected of being allergic to study drugs;
15. Patients with other organ dysfunction who are expected to be unable to tolerate general anesthesia or hepatectomy;
16. Other conditions in which the investigators deem the patients unsuitable for the clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response: Objective response rate (assessed based on mRECIST criteria) | Up to approximately 36 months
  Proportion of patients who achieve pre-defined tumor volume reduction and can maintain the minimum time limit, as the sum of complete response (CR) and partial response (PR) ratios (assessed based on mRECIST criteria)

SECONDARY OUTCOMES:
Tumor response: Objective response rate (assessed based on RECIST1.1 criteria) | Up to approximately 36 months
  Proportion of patients who achieve pre-defined tumor volume reduction and can maintain the minimum time limit, as the sum of complete response (CR) and partial response (PR) ratios (assessed based on RECIST1.1 criteria)
Overall survival (OS) | Up to approximately 36 months
  Time period from the patient's enrollment to death due to any cause.
Progression-free survival (PFS) | Up to approximately 36 months
  Time period from the patient's enrollment to the event of tumor progression or death.
Percentage of patients who can receive resection. | Up to approximately 36 months
  Percentage of patients who can receive resection.
Adverse Events as assessed by CTCAE 5.0 criteria | Up to approximately 36 months
  the main evaluation includes surgery-related adverse events, adverse events (AE), Serious adverse events (SAE), vital signs, physical examination, and laboratory examination. The severity of adverse events will be evaluated according to the NCI CTCAE 5.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No